CLINICAL TRIAL: NCT05653492
Title: Safety, Feasibility, and Tolerability of Sulforaphane in Children with CKD
Brief Title: Safety, Feasibility, and Tolerability of Sulforaphane in Children with Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Rebecca Levy, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007450
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Kidney Disease
MeSH Terms: interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): 30-50 lbs; 1 tablet (30mg/d) 50-70 lbs; 2 tablets (60mg/d) 70-90 lbs; 3 tablets (90mg/d) >90 lbs; 4 tablets (120 mg/d)
  Interventions: Drug: Sulforaphane
- Group 2 (Active Comparator): 30-50 lbs; 1 tablet (30mg/d) 50-70 lbs; 1 tablet (30mg/d) 70-90 lbs; 2 tablets (60mg/d) >90 lbs; 2 tablets (60 mg/d)
  Interventions: Drug: Sulforaphane
- Group 3 (Active Comparator): 30-50 lbs; 1 tablet (30mg/d) 50-70 lbs; 1 tablet (30mg/d) 70-90 lbs; 1 tablet (30mg/d) >90 lbs; 1 tablet (30 mg/d)
  Interventions: Drug: Sulforaphane

INTERVENTIONS:
Drug: Sulforaphane — Dosing study one to four 30 mg/d tablets depending on weight

SUMMARY:
This purpose of this study is to investigate potential new therapeutics in pediatric chronic kidney disease (CKD). The specific aims are to identify safe dosing and tolerability of sulforaphane (SFN) supplementation in children with moderate and advanced CKD. Secondary objectives will include preliminary exploration of changes in oxidative and inflammatory biomarkers in response to SFN supplementation in this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic of kidney disease
* have eGFR 20-59 mL/min/1.73m2 at the time of enrollment
* parents must be able to provide consent

Exclusion Criteria:

* weight <30 kg
* cancer or HIV diagnosis
* history of solid organ transplantation (including kidney transplant)
* structural heart disease
* currently pregnant or plan to become pregnant
* life expectancy is less than one year
* Patients will also be excluded if they are currently taking anticoagulants, immunosuppression, or chemotherapeutics

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mean half life of drug in blood | 8 hours
mean maximum concentration of drug in blood | 8 hours
mean area under the curve of drug concentration in blood | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No